CLINICAL TRIAL: NCT00734734
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of FLUAD® Surface Antigen, Inactivated, Adjuvanted With MF59C.1 Influenza Vaccine, Formulation 2008-2009, When Administered to Elderly Subjects
Brief Title: Safety and Immunogenicity of Surface Antigen, Inactivated, Adjuvanted With MF59C.1 Influenza Vaccine, Formulation 2008-2009
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70P7S; 2008-001047-19
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Interpandemic Influenza
Keywords: Prophylaxis of Influenza; Influenza Vaccines; MF59C.1
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — 1 single intramuscular dose of influenza vaccine, 2008/2009 NH formulation

SUMMARY:
Trial for annual approval of interpandemic influenza vaccines

ELIGIBILITY:
Key Inclusion Criteria:

* 65 years of age or older
* Mentally competent
* Willing and able to give written informed consent prior to study entry
* Able to comply with all the study requirements
* In general good health

Key Exclusion Criteria:

* Any serious chronic or acute disease
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g. to ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate);
* Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age)
* Receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study; suspected or known HIV infection or HIV-related disease
* A bleeding diathesis or condition associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject
* Within the past 12 months, they have received more than one injection of influenza vaccine
* Within the past 6 months, participants had laboratory confirmed influenza disease; received influenza vaccine
* Within the past 4 weeks participants had received another vaccine; any investigational agent
* An acute exacerbation of a COPD (chronic obstructive pulmonary disease) within the past 14 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (2):
- Italy (2):
  - Ufficio Igiene e Sanità Pubblica di Lanciano, ASL Lanciano - Vasto, sede legale, Lanciano
  - Pianiga Distretto n. 2 - Area Sud - Azienda ULSS 13 Mirano -Via Nazionale 48, Pianiga

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 64 participants ≥65 years of age were enrolled at 2 sites in Italy.
Pre-assignment Details: Blood samples for the determination of antibody titers were drawn on Day 0 prior to vaccination.
Groups:
- FLUAD: Participants received a single intramuscular (IM) 0.5 milliliter (mL) dose of FLUAD, a trivalent subunit inactivated adjuvanted with MF59C.1 influenza vaccine recommended for the NH 2008/2009 influenza season into the deltoid region of the non-dominant arm on Day 0 and were assessed until Day 21.
Period: Overall Study
Arm/Group | FLUAD
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was defined as all participants who were enrolled.
Groups:
- FLUAD: Participants received a single IM 0.5 mL dose of FLUAD, a trivalent subunit inactivated adjuvanted with MF59C.1 influenza vaccine recommended for the NH 2008/2009 influenza season into the deltoid region of the non-dominant arm on Day 0 and were assessed until Day 21.
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Seroconversion or Significant Increase in Single Radial Hemolysis (SRH) Area Against Each of Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants who achieved seroconversion or significant increase in single radial hemolysis (SRH) area, against each of the three vaccine strains, three weeks after vaccination (day 21), evaluated using SRH assay.
  Seroconversion: proportion of participants with negative pre-vaccination serum and a post-vaccination serum area ≥ 25 mm2. Significant increase: proportion of participants with at least a 50% increase in area from positive pre-vaccination serum. Seroconversion or significant increase: proportion of participants with either seroconversion or significant increase.
  The European (Committee for Medicinal Products for Human Use [CHMP]) criterion is met, if percentage of participants achieving seroconversion or significant increase in SRH area is 30% (≥65 years).
Time Frame: day 21
Population: Per protocol (PP) analysis set included all enrolled participants who had received the relevant dose of vaccine correctly on Day 0, provided evaluable serum samples with the relevant time windows, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Percentage of participants
  A/H1N1 | 38 [26 to 50]
  A/H3N2 | 55 [42 to 67]
  B | 42 [30 to 55]

2. Primary Outcome: Geometric Mean Ratio of Participants Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Geometric mean ratio (GMR) of participants was calculated as the ratio of post-vaccination to pre-vaccination SRH geometric mean areas (GMAs), directed against each of the three vaccine strains, three weeks after FLUAD vaccination (day 21).
  The CHMP criterion was met if the geometric mean increase (GMR, day 21/day 0) in SRH antibody area is >2.0 (≥65 years).
Time Frame: day 21
Population: Analysis was done using PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Ratio
  A/H1N1 | 1.87 [1.5 to 2.33]
  A/H3N2 | 3.74 [2.73 to 5.11]
  B | 2.38 [1.81 to 3.13]

3. Primary Outcome: Percentage of Participants Who Achieved SRH Area ≥25mm2 Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants achieving SRH area ≥25 mm2 against each of the three vaccine strains at baseline (day 0) and three weeks after FLUAD vaccination (day 21).
  This criterion is met according to CHMP guideline if percentage of participants achieving SRH area ≥25 mm2 is 60% (≥65 years).
Time Frame: day 21
Population: Analysis was done using PP set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Percentage of participants
  A/H1N1 | 89 [79 to 95]
  A/H3N2 | 75 [63 to 85]
  B | 80 [68 to 89]

4. Primary Outcome: Number of Participants Who Reported Solicited Local and Systemic Reactions
Description: Safety was assessed for participants who reported solicited local and systemic reactions from day 0 up to and including day 3 after the FLUAD vaccination.
Time Frame: 0 to 3 days post-vaccination
Population: Analysis was done using the safety dataset; participants in the exposed population who provided post-vaccination safety data.
Measure: Number; unit: Number of participants
Groups:
- FLUAD: Participants received a single IM 0.5 mL dose of FLUAD, a trivalent subunit inactivated adjuvanted with MF59C.1 influenza vaccine recommended for the NH 2008/2009 influenza season into the deltoid region of the non-dominant arm on Day 0 and were assessed until Day 3.
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Number of participants
  Injection site ecchymosis (N= 59) | 0
  Injection site erythema (N= 64) | 10
  Injection site induration (N= 64) | 2
  Injection site swelling (N= 59) | 0
  Injection site pain (N= 64) | 11
  Chills shivering (N= 64) | 0
  Malaise (N= 64) | 0
  Myalgia (N= 64) | 1
  Arthralgia (N= 64) | 0
  Headache (N= 64) | 2
  Sweating (N= 64) | 1
  Fatigue (N= 64) | 2
  Fever (≥38°C) (N= 64) | 0

ADVERSE EVENTS:
Time Frame: From Day 0 through Day 21.
Description: Adverse events other than local and systemic reactions or solicited reactions lasting longer than 3 days after vaccination were documented during the study period. Analysis was done using the safety dataset; participants in the exposed population who provided post-vaccination safety data.
Arm/Group | FLUAD
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 4/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUAD (N=64)
Induration (General disorders) | 1
Injection site erythema (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.